CLINICAL TRIAL: NCT07150039
Title: Immediate Effects of a Myofascial Diaphragm Release Technique on Thoracic Mobility and Chest Expansion in Competitive Brazilian Jiu Jitsu Athletes. A Randomized Crossover Study.
Brief Title: 20 Competitive Athletes of Brazilian Jiu Jitsu Where Randomly Assigned in a Myofascial Diaphragm Release Technique or a Sham Technique in Order to Investigate the Immediate Effects of Thoracic Mobility and Chest Expansion
Acronym: Myofascial Rx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evdokia Billis (Other)
Responsible Party: Sponsor-Investigator, Evdokia Billis, Professor in Physiotherapy, Laboratory of Clinical Physiotherapy and Research, Department of Physiotherapy, University of Patras, University of Patras
Organization: University of Patras (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Myofascial technique on BJJ
Record Dates: First submitted 2025-07-19; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Competitive Atheletes of Brazilian Jiu Jitsu
Keywords: manual therapy; myofascial reslease technique; diaphragm technique; spinal flexibility; atheletes; diaphragm myofascial release techique

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release intervention arm (Experimental): This myofascial technique was a manual hterapy treatment technique performed in sitting. With this technique, the athlete slightly bends his/her torso in order to relax the abdominal wall and breathes calmly and deeply . The therapist is behind the athlete holding his/her lower ribs, and during exhalation the therapist directs his hands caudally. This steady but gentle 'traction' is maintained throughout the breathing cycles for 4-5 minutes.
  Interventions: Other: Manual therapy intervention (Chaitow's myofascial diaphragm release)
- Sham intervention arm (Sham Comparator): With this technique (also performed in sitting), the therapist stood behind the athlete touching the outside of the person's lower ribs without folding his or her fingers or applying any pressure. The athlete is verbally instructed, after fully exhaling the air in their lungs to take deep breaths opening his/her ribs as much as he/she can whistle the therapist's hands follow the movement (without applying any manual pressure or traction). The procedure here also lasted for 4-5 minutes.
  Interventions: Other: Sham Comparison

INTERVENTIONS:
Other: Manual therapy intervention (Chaitow's myofascial diaphragm release) — Participants were given a myofascial release technique from a seated position, as described by Chaitow. With this technique, the athlete slightly bends his/her torso in order to relax the abdominal wall and breathes calmly and deeply (Figure 2). The therapist is behind the athlete holding his/her lower ribs, and during exhalation the therapist directs his hands caudally. This steady but gentle 'traction' is maintained throughout the breathing cycles for 4-5 minutes.
  Arms: Myofascial release intervention arm
Other: Sham Comparison — With this sham comparator technique, the therapist stood behind the athlete (who was sitting) touching the outside of the person's lower ribs without folding his or her fingers or applying any pressure. The athlete is verbally instructed, after fully exhaling the air in their lungs to take deep breaths opening his/her ribs as much as he/she can whistle the therapist's hands follow the movement (without applying any manual pressure or traction). The procedure here also lasted for 4-5 minutes
  Arms: Sham intervention arm

SUMMARY:
Thoracic injuries, in high level competitive Brazilian jiu jitsu (BJJ) athletes occupied a significant percentage of all musculoskeletal injuries in this population. Important factors for reducing injury rates are suggested to be spine and thoracic flexibility, which assist athletes in performing offensive/defensive techniques. The diaphragm, as one of the main thoracic and breathing muscles, appears to affect spinal flexibility and chest expansion. Thus, this study's objective was to investigate the immediate effects of a myofascial release technique of the diaphragm on chest mobility (expansion) and spinal range of movement (ROM) in BJJ athletes.

DETAILED DESCRIPTION:
In order to be assesed the immediate effects of a myofascial release technique on diaphragm, competitive BJJ athletes were subjected to a diaphragmatic release technique and to a sham breathing technique, in random order, across a two-week interval with outcome measures involving thoracic flexion/extension ROM, chest expansion, finger-to-floor (FTF) test and Modified-modified Schober's test (MMST).

ELIGIBILITY:
Inclusion Criteria:

* adult athletes up to 50 years old, with at least three years of experience in athletic BJJ competitions and participate in training sessions at least three times a week without interruption during the last year.

Exclusion Criteria:

* Athletes having sustained spinal or rib fractures in the last year or being suffering from chronic diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Chest expansion measurement as assesed by tape measure | Before and immediately after the intervention
  Chest expansion was measured in centimeters with a tape measure at two thoracic levels. For the upper chest, the anatomical landmarks used were T5 spinous process, the midline of the clavicle and the third intercostal space. For the lower chest, T10 spinous process and the xiphoid process were used.

SECONDARY OUTCOMES:
mobility of the thoracolumbar region as assesed by the Modified-modified Schober's test (MMST) | Before and immediately acfter the intervention
  The Modified-modified Schober's test (MMST) was used to measure the mobility of the lumbar/thoracolumbar region in centimeters (cm). The physiotherapist marked the midpoint between the posterior superior iliac spines on the athlete and a line was drawn 15 cm above this point with a dermatographic pen. The distance between the two marked points was measured in upright position. Then, the athlete bended forward as far as possible with knees extended, and the distance between the two marked points was measured again in flexion. The difference between the initial and final measurements in centimeters (cm) represented the lumbar/thoracolumbar total mobility
goniometry of the thoracic flexion and extension range of movement as assessed by buble inclinometers | Before and immediately after the intervention
  Two circular bubble inclinometers (goniometers) were used which calculated the range of motion in degrees. Before the measurements, the levels C7/T1 and T12/L1 were identified by palpation and marked on the athlete's body with a dermatographic pen, to point the beginning and end of the thoracic spine. The two inclinometers were then firmly placed at each point with the athlete simulating an upright posture and waited until the inclinometers calibrated to zero. The subject was then asked to bend forward with legs extended, whistle the examiner maintained the inclinometers in perpendicular contact with the marked thoracic points for recording the degree of flexion. To calculate the total thoracic flexion ROM, the A7/T1 inclinometer measurement in degrees was subtracted from that of the T12/L1 level. The same procedure was performed for extension.
overall mobility of the posterior kinetic chain as assesed by the Fingertip-to-Floor (FTF) test | Before and immediately after the intervention
  To assess the overall mobility of the posterior kinetic chain, in the FTF test the subject stood upright on a 20 cm platform with the feet together. He/She was asked to bend forward as far as he/she could while keeping knees parallel and extended with hands and fingers together in full extension. The distance between the tip of the middle finger of the right hand with the ground was measured with a tape measure in centimeters (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, Physiotherapy, Principal Investigator — University of Patras
Locations (1):
- Laboratory of Clinical Physiotherapy and Research (CPR lab), Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Yes
Happy to share primary outcome's data